CLINICAL TRIAL: NCT03037047
Title: Efficacy and Safety of Salvianolate Injection in Elderly Patients With Unstable Angina Pectoris: a Parallel, Double Blind, Randomized, Controlled, Multi-center Trial.
Brief Title: Efficacy and Safety of Salvianolate Injection in Elderly Patients With Unstable Angina Pectoris
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Valley Group of China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GV-MD-CT201601
Record Dates: First submitted 2017-01-20; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Unstable Angina
MeSH Terms: conditions — Angina, Unstable | interventions — Sodium Chloride; Saline Solution; salvianolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): patients will be treated by 0.9% sodium chloride injection on the basis of conventional therapy for 14 days.
  Interventions: Drug: 0.9% Sodium Chloride Injection
- Experimental group (Experimental): patients will be treated by salvianolate injection on the basis of conventional therapy for 14 days.
  Interventions: Drug: salvianolate injection

INTERVENTIONS:
Drug: 0.9% Sodium Chloride Injection — Patients will treated with 0.9% Sodium Chloride Injection on the basis of conventional therapy for 14 days.
  Other Names: Normal saline
  Arms: Control group
Drug: salvianolate injection — Patients will treated with salvianolate injection on the basis of conventional therapy for 14 days.
  Other Names: Salvianolate
  Arms: Experimental group

SUMMARY:
This parallel, double blind, randomized, controlled, multi-center study will evaluate the efficacy and safety of salvianolate injection in elderly patients with unstable angina pectoris.

DETAILED DESCRIPTION:
This parallel, double blind, randomized, controlled, multi-center study will evaluate the efficacy and safety of salvianolate injection in elderly patients with unstable angina pectoris. Patients will treated with or without salvianolate injection on the basis of conventional therapy for 14 days. The primary measures of effectiveness include the change from baseline to the end of treatment in the angina scores.(Angina score table :sum of 4 items), the variation of EKG (level of the S-T segment)., Additional measures of effectiveness include the change from baseline to the end of the treatment in the Seattle Angina Questionnaire(SAQ),EuroQol-5 Dimensions(EQ-5D) will be performed throughout the study. Patients who complete the double-blind portion of the study will be followed up 28 days. Effectiveness will be assessed at 7 days, 14 days and 28 days. Safety evaluations (incidence of adverse events,, physical examinations, laboratory tests) will be performed at at 7 days, 14 days and 28 days of the study.

ELIGIBILITY:
inclusion criteria

1. Patient in line with 1979 WHO diagnostic criteria for UA
2. Ages eligible for study: 60-85years (adult,senior)
3. Traditional Chinese medicine for CHD treatment should be stopped at least 1 week;take CHD drugs standardly
4. Participates give written informed consent

exclusion criteria

1. NSTE-ACS caused by non atherosclerotic disease
2. Angina pectoris caused by violent activities, fever, tachycardia, high adrenergic state, mental stress, lack of sleep, eating too full, left ventricular load increased (hypertension, aortic stenosis)
3. Angina pectoris caused byanemia, methemoglobinemia and hypoxemia
4. Abnormal thyroid function
5. Poorly controlled hypertension (systolic pressure ≥160mmHg or diastolic blood pressure ≥100mmHg)
6. Severe cardiopulmonary dysfunction
7. Severe arrhythmia (atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia, sinus bradycardia (heart rate < 55),complete left bundle branch block
8. Combined liver and kidney and hematopoietic system and other serious diseases, liver function (ALT, AST) 3 times higher than the upper limit of normal renal function, creatinine clearance rate (CrCl) less than 30 ml/min/1.73m2
9. Recent 4 weeks underwent surgery and bleeding tendency
10. Poor compliance
11. At the same time in other clinical researches
12. Allergic constitution

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
symptom of angina pectoris | up to 14 days

SECONDARY OUTCOMES:
Seattle angina scale score | up to 28 days
EQ-5D health scale | up to 28 days
thrombolysis in myocardial infarction risk score | up to 28 days
Incidence of cardiovascular and cerebrovascular events | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, doctor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospita, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cui H, Li XY, Gao XW, Lu X, Wu XP, Wang XF, Zheng XQ, Huang K, Liu F, Luo Z, Yuan HS, Sun G, Kong J, Du XH, Zheng J, Liu HY, Zhang WJ. A Prospective Randomized Multicenter Controlled Trial on Salvianolate for Treatment of Unstable Angina Pectoris in A Chinese Elderly Population. Chin J Integr Med. 2019 Oct;25(10):728-735. doi: 10.1007/s11655-019-2710-x. Epub 2019 Nov 28. PMID 31782009